CLINICAL TRIAL: NCT04837937
Title: Negotiation Training to Optimize Caregiver Communication in Alzheimer's Disease
Brief Title: Negotiation Training for Caregiver Communication in AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lee Lindquist, Associate Professor of Medicine, Chief - Geriatrics, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: R01AG068421-01 (NIH); 1R01AG068421-01 (NIH)
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Cognitive Impairment
Keywords: Family caregiver; Negotiation; Dispute resolution; Conflict communication
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Negotiating

STUDY DESIGN:
Intervention Model Description: The randomized controlled clinical trial has a full factorial testing 3 components at 2 levels each (on and off).
  Individuals will be randomized to 1 of 8 experimental conditions. Participants can be assigned to intervention ("Yes") or control ("No") conditions for each component. All participants will receive a "caregiver-patient" negotiation exercise so that no participant gets an inactive placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise. All participants will complete this exercise; it will serve as the constant.
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]
- Condition 2 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Patient [Advanced]' ' conflict negotiation/dispute resolution exercise
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]; Behavioral: Caregiver vs. Patient [Advanced]
- Condition 3 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]; Behavioral: Caregiver vs. Physician
- Condition 4 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Patient [Advanced]' conflict negotiation/dispute resolution exercise
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]; Behavioral: Caregiver vs. Physician; Behavioral: Caregiver vs. Patient [Advanced]
- Condition 5 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]; Behavioral: Caregiver vs. Caregiver
- Condition 6 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Patient [Advanced]' conflict negotiation/dispute resolution exercise
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]; Behavioral: Caregiver vs. Caregiver; Behavioral: Caregiver vs. Patient [Advanced]
- Condition 7 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]; Behavioral: Caregiver vs. Caregiver; Behavioral: Caregiver vs. Physician
- Condition 8 (Experimental): (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise; (4) 'Caregiver vs. Patient [Advanced]' conflict negotiation/dispute resolution exercise
  Interventions: Behavioral: Caregiver vs. Patient [Beginner]; Behavioral: Caregiver vs. Caregiver; Behavioral: Caregiver vs. Physician; Behavioral: Caregiver vs. Patient [Advanced]

INTERVENTIONS:
Behavioral: Caregiver vs. Patient [Beginner] — Participants will be assigned a 'Caregiver vs. Patient' [Beginner] online negotiation exercise. All participants will complete this exercise, so it will serve as the constant.
Behavioral: Caregiver vs. Caregiver — Participants will be assigned a 'Caregiver vs. Caregiver' online negotiation exercise.
  Arms: Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Caregiver vs. Physician — Participants will be assigned a 'Caregiver vs. Physician' online negotiation exercise.
  Arms: Condition 3; Condition 4; Condition 7; Condition 8
Behavioral: Caregiver vs. Patient [Advanced] — Participants will be assigned a 'Caregiver vs. Patient [Difficult]' online negotiation exercise. This exercise is "advanced" compared to the constant since it involves negotiating more than one conflict.
  Arms: Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
The purpose of this study is to design a Negotiation and Dispute Resolution (NDR) training intervention to improve communication and address resolution of conflicts that family caregivers of patients with cognitive impairment and/or Alzheimer's Disease (AD) frequently experience.

DETAILED DESCRIPTION:
The goal of this study is to design a Negotiation and Dispute Resolution (NDR) training intervention to improve communication and address resolution of conflicts that family caregivers of patients with cognitive impairment and/or Alzheimer's Disease (AD) frequently experience. Specifically this study will:

Aim 1: Employ a caregiver (user)-centered design approach to modify and tailor a negotiations and dispute resolution (NDR) training intervention to support communication skills of family caregivers of adults with AD.

Aim 2: Utilizing Multiphase Optimization Strategy (MOST), conduct a randomized controlled trial of the NDR intervention that targets better communication between caregivers and health teams to determine the feasibility of delivering the intervention, and derive estimates of the effect of 3 intervention components on changes in patient-centered outcomes at post-intervention and follow-up.

Exploratory Aim 3: Explore if intervention components (lectures/exercises) interact to change communication between caregivers and health care teams at post-intervention and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Speak/read English;
* Currently provide care-giving support (e.g. emotional, social, physical, task-related) to an adult over the age of 65;
* Currently provide care-giving support at least 1 hour per week (e.g. may include grocery shopping, scheduling appointments, and transportation);
* Currently involved in any decision-making related to the healthcare and support of this adult over the age of 65;
* Score >2 on the 8-item Informant Interview to Differentiate Aging and Dementia (AD8);
* Access to and the ability to use the internet to complete a series of online activities; and
* Have a valid email address or the willingness to create one to access during the study

Exclusion Criteria:

* Less than 21 years old
* Unable to speak and read English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olvera C, Ramirez-Zohfeld V, Murawski A, Pfammatter AF, Lindquist LA. Evaluating a negotiation training program for family caregivers of older people using a Multiphase Optimization Strategy (MOST) design and protocol. Contemp Clin Trials Commun. 2026 Jan 12;49:101596. doi: 10.1016/j.conctc.2026.101596. eCollection 2026 Feb. PMID 41607873

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants consented but were not randomized to a condition. One of these participants did not complete baseline intake and was not randomized to a treatment. The other participant did complete baseline intake but did not complete the study phase which assigns participants to a condition (a unique hyperlink which assigns condition and treatment materials when opened- this participant did not open their link).
Groups:
- Universal: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise. All participants will complete this exercise; it will serve as the constant.
- Older Adult: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Patient [Advanced]' ' conflict negotiation/dispute resolution exercise
- Physician: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise
- Physician/OA: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Patient [Advanced]' conflict negotiation/dispute resolution exercise
- Sister: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise
- Sister/OA: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Patient [Advanced]' conflict negotiation/dispute resolution exercise
- Sister/Physician: (1) 'Caregiver vs. Patient [Beginner]' negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise
- Sister/Physician/OA: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise; (2) 'Caregiver vs. Caregiver' conflict negotiation/dispute resolution exercise; (3) 'Caregiver vs. Physician' conflict negotiation/dispute resolution exercise; (4) 'Caregiver vs. Patient [Advanced]' conflict negotiation/dispute resolution exercise
Period: Overall Study
Arm/Group | Universal | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Started | 15 | 17 | 16 | 16 | 17 | 16 | 17 | 17
Completed | 15 | 15 | 15 | 15 | 16 | 15 | 17 | 16
Not Completed | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Universal Only: (1) 'Caregiver vs. Patient [Beginner]' conflict negotiation/dispute resolution exercise. All participants will complete this exercise; it will serve as the constant.
- Total: Total of all reporting groups
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA | Total
Number analyzed (Participants) | 15 | 17 | 16 | 16 | 17 | 16 | 17 | 17 | 131
Age, Continuous [Mean (Full Range); unit: Years] | 58.33 [52 to 67] | 55.71 [27 to 75] | 56.81 [29 to 76] | 55.56 [28 to 73] | 48.76 [27 to 71] | 51.44 [21 to 78] | 53.23 [21 to 75] | 51.59 [25 to 79] | 53.64 [21 to 79]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 12 | 14 | 13 | 12 | 11 | 13 | 15 | 11 | 101
  Sex/Gender: Male | 3 | 3 | 3 | 4 | 6 | 3 | 2 | 5 | 29
  Sex/Gender: Non-Binary | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 1 | 0 | 2 | 0 | 3 | 10
  Not Hispanic or Latino | 14 | 16 | 11 | 14 | 16 | 12 | 15 | 13 | 111
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 5 | 5 | 5 | 4 | 6 | 3 | 5 | 6 | 39
  White | 9 | 11 | 9 | 9 | 10 | 11 | 10 | 11 | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 5
Positive Affect and Well-Being [Mean (Standard Deviation); unit: T-Score] — Positive Affect and Well-Being as measured at baseline by Neuro-QoL Positive Affect and Well Being scale. Population mean T-Score is 50 with an SD of 10. Higher scores on the scale represent better self-reported health (i.e. higher score=more positive affect and well being).
  T-Score | 55.41 (4.07) | 56.22 (6.97) | 55.5 (6.84) | 56.83 (7.23) | 54.2 (5.87) | 52.83 (5.66) | 54.86 (4.84) | 53.9 (5.92) | 54.96 (5.98)

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuro-QoL Positive Affect and Well-Being Score
Description: Caregiver well-being as measured by the Positive Affect and Well-being scale for the Neurology Quality of Life (Neuro-QOL). The measure is a 9-item panel rating how caregivers experience feelings of positive affect and well-being. Responses are Likert scales, scored 1-5, Never (1), Rarely (2), Sometimes (3), Often (4), Always (5). Responses are summed for a final score and converted to a t-score per Neuro-QoL manual scoring conventions. Population mean T-Score is 50 and SD is 10. Higher scores indicate higher levels of Positive Affect and Well-Being. Positive change represents an increase in positive affect/well-being, and negative change represents a decrease.
Time Frame: Baseline (pre-intervention) and 1 Month Post-intervention
Population: All participants with available data at baseline and 1 month post-intervention assessments were analyzed.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 17 | 16 | 16 | 17 | 16 | 17 | 17
T-Score
  Baseline (Pre-Intervention) | 55.41 (4.07) | 56.22 (6.94) | 55.51 (6.84) | 56.83 (7.23) | 54.2 (5.87) | 52.83 (5.66) | 54.86 (4.84) | 53.9 (5.92)
  1 month Post Intervention: number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
  1 month Post Intervention | 54.39 (5.59) | 55.74 (4.82) | 53.66 (6.22) | 53.76 (6.84) | 54.51 (6.51) | 53.01 (5.19) | 54.69 (4.86) | 54.45 (5.28)
Statistical Analysis 1: Comparison: Physician; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "physician" treatment arm; Test type: Superiority; p = .7695, Mixed Models Analysis — Alpha for significance=0.05 for all tests; Mean Difference (Final Values) = .1491, 95% CI [-.856 to 1.15], Standard Error of Mean .51
Statistical Analysis 2: Comparison: Sister; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "sister" treatment arm; Test type: Superiority; p = .0878, Mixed Models Analysis — ALPHA=0.05; Mean Difference (Final Values) = -.87, 95% CI [-1.88 to .13], Standard Error of Mean .5077
Statistical Analysis 3: Comparison: Sister/Physician; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "sister/physician" treatment arm; Test type: Superiority; p = .635, Mixed Models Analysis — ALPHA=0.05; Mean Difference (Final Values) = .2414, 95% CI [-.76 to 1.25], Standard Error of Mean .5077
Statistical Analysis 4: Comparison: Older Adult; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "older adult" treatment arm; Test type: Superiority; p = .897, Mixed Models Analysis — ALPHA=0.05; Mean Difference (Final Values) = -.06574, 95% CI [-1.0709 to .9394], Standard Error of Mean .5077
Statistical Analysis 5: Comparison: Physician/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "physician/older adult" treatment arm; Test type: Superiority; p = .9823, Mixed Models Analysis — ALPHA=0.05; Mean Difference (Final Values) = -.01126, 95% CI [-1.0164 to .9939], Standard Error of Mean .5077
Statistical Analysis 6: Comparison: Sister/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "sister/older adult" treatment arm; Test type: Superiority; p = .3337, Mixed Models Analysis — ALPHA=0.05; Mean Difference (Final Values) = -.4928, 95% CI [-1.4979 to .5124], Standard Error of Mean .5077
Statistical Analysis 7: Comparison: Sister/Physician/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "sister/older adult/physician" treatment arm; Test type: Superiority; p = .694, Mixed Models Analysis — ALPHA=0.05; Mean Difference (Final Values) = .2002, 95% CI [-.8049 to 1.2054], Standard Error of Mean .5077
Statistical Analysis 8: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the intercept (all tx=0); Test type: Superiority; p < .0001, Mixed Models Analysis — this is the Intercept value for the GLMM evaluating all combinations of treatment and time- in other words, this is the mean well-being t-score across all combinations of tx and time. Estimates in these analyses are deviations from this intercept; Actual Intercept value = 54.9056, 95% CI [53.9003 to 55.9109], Standard Error of Mean .5077
Statistical Analysis 9: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This test evaluates the effect of time (measured as weeks since baseline); Test type: Superiority; p = .1152, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = -.05579, 95% CI [-.1254 to .01383], Standard Error of Mean .03516
Statistical Analysis 10: Comparison: Physician; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "Physician" treatment arm*time; Test type: Superiority; p = .3555, Mixed Models Analysis; Mean Difference (Final Values) = -.03261, 95% CI [-.1022 to .03699], Standard Error of Mean .03516
Statistical Analysis 11: Comparison: Sister; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "sister" treatment arm*time; Test type: Superiority; p = .0546, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = .06825, 95% CI [-.00136 to .1379], Standard Error of Mean .03516
Statistical Analysis 12: Comparison: Sister/Physician; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "Sister/Physician" treatment arm*time; Test type: Superiority; p = .4616, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = .02597, 95% CI [-.04364 to .09557], Standard Error of Mean .03516
Statistical Analysis 13: Comparison: Older Adult; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "Older Adult" treatment arm*time; Test type: Superiority; p = .1592, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = .0498, 95% CI [-.0198 to .1194], Standard Error of Mean .03516
Statistical Analysis 14: Comparison: Physician/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "Physician/Older Adult" treatment arm*time; Test type: Superiority; p = .4899, Mixed Models Analysis; Mean Difference (Final Values) = -.02435, 95% CI [-.09396 to .04526], Standard Error of Mean .03516
Statistical Analysis 15: Comparison: Sister/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "sister/older adult" treatment arm*time; Test type: Superiority; p = .9842, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = .000697, 95% CI [-.06891 to .0703], Standard Error of Mean .03516
Statistical Analysis 16: Comparison: Sister/Physician/OA; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing all levels and combinations of treatments and time as fixed effects, controlling for repeated assessments within-subjects, for effect on the outcome of change in Neuro-QoL positive affect and well being score. This result is for the "Sister/Older Adult/Physician" treatment arm*time; Test type: Superiority; p = .7217, Mixed Models Analysis — alpha=0.05; Mean Difference (Final Values) = -.01255, 95% CI [-.08216 to .05705], Standard Error of Mean .03516

2. Secondary Outcome: Change in PROMIS Anxiety Score
Description: The PROMIS Adult Emotional Distress-Anxiety scale measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), and hyper-arousal (tension, nervousness, restlessness) in respondents during the past 7 days. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always). We deployed the four item short form, with scores ranging from 4-20, with higher scores indicating greater severity of anxiety. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. We calculate change in T-Score from baseline to one month per participant and take the mean of those observations to produce mean change in T-score by condition.
Time Frame: 1 months post-baseline
Population: All participants who were randomized and completed the 1 month post-intervention assessment are included in the change analysis (n=125).
Measure: Mean (Standard Deviation); unit: Change in T-Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
Change in T-Score | .52 (5.43) | -1.81 (7.43) | -.81 (8.11) | -.04 (6.87) | -1.06 (4.88) | -.52 (4.37) | 1.74 (5.09) | -4.11 (8.80)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA- analytic variable is change in PROMIS Anxiety score from baseline to T3. Test is a paired T-Test; Test type: Superiority; p = .21, 2-sided paired t-Test — Threshold for statistical significance was alpha=0.05; Mean Difference (Final Values) = -.74, 95% CI [-1.90 to .42], Standard Deviation 6.55

3. Secondary Outcome: Change in Zarit Caregiver Burden Score
Description: The Zarit Burden Interview, a popular caregiver self-report measure used by many aging agencies, originated as a 29-item questionnaire (Zarit, Reever & Bach-Peterson, 1980). The revised version contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). The total score range is 0 to 88. Increasing scores indicate increasing burden.
  Scores were measured at baseline and at 1 month post-intervention and a change score was computed for each participant. These change scores are averaged to produce the by-condition mean change in burden score. Positive results indicate an increase in burden, and negative results indicate a decrease in burden.
Time Frame: 1 month post-baseline
Population: All participants with data available at 1 months post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in Burden Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
Change in Burden Score | -.07 (7.69) | -3.21 (11.22) | -9.6 (12.05) | -.44 (12.62) | -3.35 (7.93) | 0 (14.35) | -2.59 (8.45) | -6.69 (14.97)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Zarit Caregiver Burden Score, Baseline to 1-month post-intervention. Test was a 2-sided dependent samples t-test; Test type: Superiority; p = .0021, 2-sided dependent sample t-test — Threshold for significance was 0.05; Mean Difference (Final Values) = -3.24, 95% CI [-5.28 to -1.20], Standard Deviation 11.54

4. Secondary Outcome: Change in PROMIS Fatigue Score
Description: The PROMIS Fatigue instruments evaluate a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. We deployed PROMIS Fatigue Form 7a, a seven item likert scale panel ranging from 1=never to 5=always. Scores range from 7-35. Higher scores indicate more fatigue. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. We calculate change in T-Score from baseline to one month per participant and take the mean of those observations to produce mean change in T-score by condition.
Time Frame: 1 month post-baseline
Population: All participants with data available at 1 months post baseline were included in the analysis.
Measure: Mean (Standard Error); unit: Change in T-Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
Change in T-Score | -2.58 (6.29) | -2.9 (8.86) | -.36 (7.43) | .08 (5.22) | -4.12 (5.88) | 3.33 (9.9) | 1.36 (5.97) | -4.26 (11.72)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA- analytic variable is change in PROMIS Fatigue score from baseline to T3. Test is a paired T-Test; Test type: Superiority; p = .10, 2-Sided Paired T Test — Alpha for statistical significance was 0.05; Mean Difference (Final Values) = -1.19, 95% CI [-2.62 to .25], Standard Deviation 8.10

5. Secondary Outcome: Change in PROMIS Short Form General Self Efficacy T Score
Description: the PROMIS General Self-Efficacy - Short Form is a four item panel which measures confidence in one's ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations. The four items are 1-5 Likert scales, 1=never, 5=always. Minimum score is a 4 and maximum is a 20. Raw Scores are converted to T scores with mean 50 and SD 10 per the PROMIS scoring manual. Higher score=greater self efficacy.
Time Frame: 1 months post-baseline
Population: All participants with data available at 1 months post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: change in T-Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
change in T-Score | -.57 (5.24) | 1.22 (11.63) | .55 (8.29) | -1.32 (6.13) | .68 (10.14) | .06 (7.57) | -2.14 (5) | 1.59 (7.74)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in PROMIS short form General Self Efficacy T-Score, baseline to one month post-intervention. Test is a 2-sided paired (dependent sample) t-test; Test type: Superiority; p = .9754, 2-sided paired (dependent sample) t-test; Mean Difference (Final Values) = .02, 95% CI [-1.36 to 1.41], Standard Deviation 7.83

6. Secondary Outcome: PROMIS Short Form Emotional Support T Score at Baseline
Description: PROMIS Emotional Support - Short Form.
  The PROMIS Emotional Support item bank assesses perceived feelings of being cared for and valued as a person; having confident relationships. The short form 6a deployed here is a 6 item likert scale panel, which assesses responses as 1=never and 5=always in response to item statements. Minimum score is a 6 and maximum is a 30. Higher scores indicate greater feelings of emotional support. The raw score is rescaled per the PROMIS scoring manual into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean.
Time Frame: Baseline Measure
Population: All individuals who received and completed the baseline assessment are included in the analysis population (N=131).
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 17 | 16 | 16 | 17 | 16 | 17 | 17
T-Score | 50.42 (9.28) | 54.93 (9.35) | 52.23 (9.77) | 52.00 (9.44) | 52.26 (10.19) | 51.68 (9.37) | 52.38 (6.62) | 50.58 (8.03)

7. Secondary Outcome: Change in PROMIS Satisfaction With Social Roles/Activities Score
Description: The PROMIS adult Satisfaction with Social Roles and Activities item bank assesses satisfaction with performing one's usual social roles and activities (e.g., "I am satisfied with my ability to participate in family activities"). Short form 8a is deployed here. This is an 8 item likert scale panel, with responses rated 1=never and 5=always. Scores range from 8 to 40. Higher scores indicate greater satisfaction with social roles and activities. The raw score is rescaled per the PROMIS scoring manual into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean.
Time Frame: 1 months post-baseline
Population: All participants with data available at 1 months post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in T Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
Change in T Score | .9 (4.7) | 2.17 (5.58) | .49 (5.55) | -1.45 (5.29) | -.09 (4.42) | -.92 (5.51) | -.55 (2.82) | .79 (5.26)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in T-Score between baseline and 1 month post-intervention. Test is a 2-sided paired t-test; Test type: Superiority; p = .77, 2-sided Paired T-Test — Threshold for significance is 0.05; Mean Difference (Final Values) = .1296, 95% CI [-.74 to 1.00], Standard Deviation 4.91

8. Secondary Outcome: Change in Neuro-QoL Caregiver Specific Anxiety Score
Description: TBI-CareQOL is a set of self-report measures within the Neuro-QoL™ measurement system that assesses the health-related quality of life (HRQOL) of caregivers of adults with traumatic brain injury (TBI). Among these is the Caregiver specific anxiety measure. This is a six item likert panel with responses rated 1=never and 5=always, for a combined score range of 6-30. Higher scores indicate greater levels of anxiety. Raw scores were rescaled per the Neuro-QoL scoring manual into T-Scores with a mean of 50 and an SD of 10. Difference between T-score at baseline and 1-month was computed for each participant to produce a change score, and these change scores are averaged to produce per condition means.
Time Frame: 1 month post-baseline
Population: All participants with data available at 1 months post baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: change in T-Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
change in T-Score | -.31 (4.12) | -2.21 (7.09) | -2.48 (6.36) | .27 (7.71) | -.37 (7.17) | .58 (6.69) | -.39 (4.33) | -1.4 (5.63)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in T-score between baseline and one month post-intervention. Test is a two-sided paired t-test; Test type: Superiority; p = .1694, two-sided paired T-Test — alpha threshold for significance was 0.05; Mean Difference (Final Values) = .7618, 95% CI [-.33 to 1.85], Standard Deviation 6.16

9. Other Pre Specified Outcome: Participant Retention Rate at 3 Months Post-baseline
Description: Percentage- numerator=# of participants who completed 3 month post-baseline assessment, denominator=# of participants randomized to a condition.
Time Frame: 3 months post-baseline
Population: 131 participants were randomized from a total 133 consented- 2 did not complete pre-randomization activities. Here we were interested in the raw number of recruited participants retained regardless of intervention received, thus all participants were considered in the analysis and group segmentation would be inappropriate for the calculation.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Randomized at Baseline: All Participants Randomized at Baseline
Arm/Group | All Participants Randomized at Baseline
Number analyzed (Participants) | 131
Participants | 124

10. Other Pre Specified Outcome: System Usability Scale Score
Description: Measuring the feasibility of the intervention by measuring the usability of the intervention as measured by the System Usability Scale (SUS), a 10-item measure of usability. SUS is a 10-item likert panel, with scores ranging from 1-5. Scores are tabulated by converting raw scores by subtracting 1 from each raw score and then summing per the scoring manual: summed score=2.5*(20+(sum of odd numbered questions)-(sum of even number questions)). The minimum and maximum values are thus 50 and 100. Higher scores indicate greater usability.
Time Frame: 2 weeks post-intervention
Population: 128 participants of 131 randomized completed the 2 weeks post-intervention assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 16 | 16 | 16 | 17 | 15 | 17 | 16
score on a scale | 68 (16) | 68 (16) | 68 (17) | 65 (12) | 73 (14) | 71 (13) | 63 (17) | 67 (19)

11. Other Pre Specified Outcome: USE Acceptability Score
Description: The USE Acceptability score measures the acceptability of the intervention, employing an 8-item panel of 1-7 Likert scale questions, with a 0 option for "not applicable". Raw score is converted to 0-100 score as follows: 2.040163*(summed raw scores - 8). Higher scores indicate greater acceptability.
Time Frame: 2 weeks post-intervention
Population: 128 of 131 randomized participants completed the post-intervention assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 16 | 16 | 16 | 17 | 15 | 17 | 16
score on a scale | 78 (11) | 73 (22) | 74 (20) | 74 (12) | 65 (23) | 80 (12) | 71 (19) | 70 (67)

12. Other Pre Specified Outcome: Exercise Completion Rate
Description: Measuring the feasibility of the intervention by assessing completion of negotiation training exercises.
Time Frame: 2 weeks post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 17 | 16 | 16 | 17 | 16 | 17 | 17
Participants | 15 | 16 | 16 | 16 | 17 | 15 | 17 | 16

13. Other Pre Specified Outcome: Change in DUTCH Conflict Handling Scores
Description: The Dutch Test for Conflict Handling measures aspects of conflict resolution pertaining to the negotiator. The DUTCH measures conflict handling in five domains: avoiding, forcing, yielding, problem solving, and compromising. Each domain is measured independently using panels of four 1-5 likert scale questions each. Domain scores thus range from 5-20, converted to 0-100 with the following formula: 6.25*(domain score-1). Intra-participant change is measured for each subdomain between baseline and 1 month and generalized to produce mean change per domain. Higher scores per domain indicate more intense conflict handling behavior in the given domain- lower scores indicate less intensity.
Time Frame: 1 month post-baseline
Population: All 125 participants who completed both the baseline and 1-month post-intervention assessments are included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in Domain Score (out of 100)
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
Change in Domain Score (out of 100)
  Change in Compromising Score | 2.08 (13.71) | 6.25 (17.68) | 2.92 (16.17) | 3.52 (18.25) | 3.31 (13.82) | 2.08 (19.72) | -2.94 (12.13) | 1.56 (20.22)
  Change in Forcing Score | -7.5 (13.19) | -9.38 (14.66) | -2.5 (18.57) | -18.36 (28.09) | -3.68 (15.63) | -9.17 (14.92) | -3.31 (14.34) | -1.56 (23.11)
  Change in Problem Solving Score | -2.08 (13.08) | 8.48 (13.56) | -6.67 (17.43) | 0 (16.93) | 4.04 (17.25) | 1.67 (14.46) | -2.57 (9.13) | -4.3 (19.06)
  Change in Yielding Score | -5.42 (13.12) | -1.79 (13.74) | -3.33 (14.54) | -1.95 (10.88) | 3.68 (11.49) | 2.5 (12.90) | 1.1 (11.32) | -4.3 (9.87)
  Change in Avoiding Score | 11.25 (19.51) | .89 (15.08) | -1.25 (17.55) | -9.38 (13.31) | -.37 (13.34) | -.83 (14.73) | -.74 (14.3) | -2.34 (19.48)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Avoiding Score (out of 100) between Baseline and 1 Month Post-Intervention; Test type: Superiority; p = .76, ANOVA — Alpha for Significance=0.05; Mean Difference (Final Values) = -.45, Standard Deviation 16.44
Statistical Analysis 2: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Compromising Score (out of 100) between Baseline and 1 Month Post-Intervention; Test type: Superiority; p = .13, ANOVA — Alpha for significance=0.05; Mean Difference (Final Values) = 2.25, Standard Deviation 16.33
Statistical Analysis 3: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Forcing Score (out of 100) between Baseline and 1 Month Post-Intervention; Test type: Superiority; p < .0001, ANOVA — Alpha for significance=0.05; Mean Difference (Final Values) = -6.85, Standard Deviation 18.76
Statistical Analysis 4: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Problem Solving Score (out of 100) between Baseline and 1 Month Post-Intervention; Test type: Superiority; p = .86, ANOVA — Alpha for Significance=0.05; Mean Difference (Final Values) = -.25, Standard Deviation 15.62
Statistical Analysis 5: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Yielding Score (out of 100) between Baseline and 1 Month Post-Intervention; Test type: Superiority; p = .32, ANOVA — Alpha for significance=0.05; Mean Difference (Final Values) = -1.1, Standard Deviation 12.30

14. Other Pre Specified Outcome: Change in Negotiation Knowledge Scores
Description: We deployed a panel of 15 questions measuring participant knowledge of negotiation techniques. The panel measures knowledge in three subdomains (identification of interests, rights, and power statements) and can also be measured in aggregate to assess knowledge across the three subdomains. Participants receive 1 point for each correct answer. All Scores, including subdomain scores, are converted to a 0/100 measure. Intraparticipant change is assessed between baseline and 1 month post-intervention. Dependent Sample T-Tests were performed on the change scores from baseline-1 month.
Time Frame: 1 months post-baseline
Population: All Participants who completed the 1 month post-intervention assessment are included.
Measure: Mean (Standard Deviation); unit: Change in Score Baseline-1 Month
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
Change in Score Baseline-1 Month
  Change in total score | 6.22 (11.94) | -1.9 (11.23) | .89 (19.82) | 8.33 (14.91) | 4.71 (9.65) | 3.11 (12.82) | 2.35 (13.11) | .42 (9.57)
  Change in Interests score | 6.67 (12.28) | 1.19 (10.26) | -1.11 (27.79) | 9.38 (21.05) | 7.84 (17.79) | 4.44 (17.21) | 4.9 (11.43) | 5.21 (15.77)
  Change in Power Score | 0 (23.15) | -3.57 (13.36) | -1.67 (25.82) | 7.81 (17.6) | 0 (17.68) | 1.67 (25.82) | -1.47 (20.67) | -1.56 (11.06)
  Change in Rights Score | 10.67 (31.95) | -4.29 (19.5) | 5.33 (22) | 7.5 (21.76) | 4.71 (16.63) | 2.67 (16.68) | 2.35 (28.18) | -3.75 (18.21)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in total Negotiation Knowledge score, Baseline 1-month. Threshold for significance was alpha=0.05; Test type: Superiority; p = .0012, ANOVA; Mean Difference (Final Values) = 3.09, Standard Deviation 13.18
Statistical Analysis 2: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Negotiation Knowledge Interests score, Baseline 1-month. Threshold for significance was alpha=0.05; Test type: Superiority; p = .0018, ANOVA — alpha=0.05; Mean Difference (Final Values) = 4.933, Standard Deviation 17.33
Statistical Analysis 3: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Negotiation Knowledge Power score, Baseline 1-month; Test type: Superiority; p = .91, ANOVA — Threshold for significance was alpha=0.05; Mean Difference (Final Values) = .2, Standard Deviation 19.69
Statistical Analysis 4: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in Negotiation Knowledge Rights score, Baseline 1-month; Test type: Superiority; p = .11, ANOVA — Threshold for significance was alpha=0.05; Mean Difference (Final Values) = 3.2, Standard Deviation 22.35

15. Other Pre Specified Outcome: Utilization Rates
Description: We deployed a survey panel of 5 yes/no questions to participants asking them about utilization of negotiation techniques in the month following the intervention. Result rates are out of 100%.
Time Frame: 1 month post-baseline
Population: 125 participants out of 131 randomized had data available at one month post-intervention. Of those, only 85 were deployed the website utilization question.
Measure: Count of Participants; unit: Participants
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 17 | 16
Participants
  In the past month, have you visited NegotiAge.com?: number analyzed (Participants) | 10 | 10 | 10 | 11 | 12 | 9 | 12 | 11
  In the past month, have you visited NegotiAge.com?: No | 4 | 7 | 7 | 4 | 5 | 5 | 5 | 4
  In the past month, have you visited NegotiAge.com?: Yes | 6 | 3 | 3 | 7 | 7 | 4 | 7 | 7
  In the past month, have you experienced any conflicts related to the care of your older adult?: No | 8 | 7 | 5 | 6 | 12 | 8 | 5 | 7
  In the past month, have you experienced any conflicts related to the care of your older adult?: Yes | 7 | 7 | 10 | 10 | 5 | 7 | 12 | 9
  In the past month, have you used anything you learned from the negotiation training activities?: No | 6 | 6 | 9 | 8 | 10 | 8 | 13 | 13
  In the past month, have you used anything you learned from the negotiation training activities?: Yes | 9 | 8 | 6 | 8 | 7 | 7 | 4 | 3
  Are there other parts of your life where you used negotiation skills gained during this study?: No | 6 | 6 | 9 | 8 | 10 | 8 | 13 | 13
  Are there other parts of your life where you used negotiation skills gained during this study?: Yes | 9 | 8 | 6 | 8 | 7 | 7 | 4 | 3
  In the past month, have you negotiated anything related to the care of your older adult?: No | 9 | 5 | 6 | 7 | 11 | 5 | 8 | 9
  In the past month, have you negotiated anything related to the care of your older adult?: Yes | 6 | 9 | 9 | 9 | 6 | 10 | 9 | 7

16. Other Pre Specified Outcome: Change In Positive and Negative Affect Schedule Scores
Description: The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point verbal frequency scale of 1 (not at all) to 5 (very much). Scores are evaluated out of 50. The ten item scales thus have score ranges from 10-50. Higher scores in a single domain indicate greater perception of that type of affect. So, higher positive affect scores=greater positive affect, and higher negative affect scores=higher negative affect. Positive change on either scale indicates an increase in that domain, and negative change on either scale indicates a decrease in that domain.
Time Frame: 1 month post-baseline
Population: All participants with data available at 1 month post-intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in Score
Arm/Group | Universal Only | Older Adult | Physician | Physician/OA | Sister | Sister/OA | Sister/Physician | Sister/Physician/OA
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 17 | 15 | 16 | 16
Change in Score
  Positive Affect Score | -.53 (2.7) | 1.21 (4.69) | 0 (5.15) | .75 (5.72) | .76 (3.98) | .2 (4.89) | .47 (4.35) | -.13 (7.11)
  Negative Affect Score | -.2 (4.06) | -2.21 (5.15) | -2.67 (5.74) | -2.19 (7.13) | -2.12 (5.05) | -1.2 (4.75) | -1.76 (6.19) | -4.19 (7.26)
Statistical Analysis 1: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA on change in negative affect score, baseline-1 month post-intervention. Test is a 2 sided dependent sample t-test; Test type: Superiority; p < .0001, 2-sided dependent sample t-test — Threshold for significance is alpha=0.05; Mean Difference (Final Values) = -2.08, 95% CI [-3.09 to -1.07], Standard Deviation 5.73
Statistical Analysis 2: Comparison: Universal Only vs Older Adult vs Physician vs Physician/OA vs Sister vs Sister/OA vs Sister/Physician vs Sister/Physician/OA; Univariate ANOVA of change in positive affect score between baseline-1 month post-intervention. Test is a 2-sided dependent sample t-test; Test type: Superiority; p = .4305, 2-sided dependent sample t-test; Mean Difference (Final Values) = .3440, 95% CI [-.52 to 1.21], Standard Deviation 4.86

ADVERSE EVENTS:
Time Frame: From Baseline enrollment (pre-intervention) until end of study (3 months post-intervention)
Description: Adverse event (AE):Any unfavorable and unintended sign or symptom temporally associated with the NDR training, regardless of whether it is considered related to intervention. Serious Adverse Event (SAE):Any AE that results in: a life-threatening situation (places the subject at immediate risk of death from the event as it occurred); death; inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant disability or incapacity.
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/16 | 0/16 | 0/17 | 0/16 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/16 | 0/16 | 0/17 | 0/16 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/16 | 0/16 | 0/17 | 0/16 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04837937/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04837937/SAP_001.pdf
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT04837937/ICF_002.pdf